CLINICAL TRIAL: NCT06423274
Title: A Comparative Analysis of the Diagnostic Outcomes of Artificial Intelligence-assisted Fundus Photography for Diabetic Retinopathy and Diabetic Macular Edema Versus Other Imaging Devices in Ophthalmology: A Controlled Trial
Brief Title: Comparing Artificial Intelligence for Assisted Diagnosis of Diabetic Retinopathy
Status: Not yet recruiting | Type: Observational
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Wu Hongkang, Director, Second Affiliated Hospital, School of Medicine, Zhejiang University
Other Study IDs: DR artificial intelligence
Record Dates: First submitted 2024-05-09; First posted 2024-05-21 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Diabetic Retinopathy; Diabetic Macular Edema
Keywords: diabetic retinopathy; diabetic macular edema; artificial intelligence
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Fluorescein Angiography; Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- artificial intelligence-assisted fundus photography: Artificial intelligence-assisted fundus photography in patients with diabetic retinopathy
  Interventions: Diagnostic Test: fundus photography
- optical coherence tomography: optical coherence tomography in patients with diabetic retinopathy
  Interventions: Diagnostic Test: optical coherence tomography
- fundus fluorescence angiography: fundus fluorescence angiography in patients with diabetic retinopathy
  Interventions: Diagnostic Test: fundus fluorescence angiography

INTERVENTIONS:
Diagnostic Test: fundus photography — using artificial intelligence to identify diabetic retinopathy using fundus photography
  Groups: artificial intelligence-assisted fundus photography
Diagnostic Test: optical coherence tomography — detect diabetic retinopathy and diabetic macular edema by optical coherence tomography
  Groups: optical coherence tomography
Diagnostic Test: fundus fluorescence angiography — detect diabetic retinopathy by fundus fluorescence angiography
  Groups: fundus fluorescence angiography

SUMMARY:
This study plans to compare the accuracy of artificial intelligence (AI)-assisted fundus images with other ophthalmic devices such as optical coherence tomography (OCT) and fundus fluorescence angiography (FFA) in the diagnosis of diabetic retinopathy and diabetic macular edema.

DETAILED DESCRIPTION:
This study plans to compare the accuracy of artificial intelligence (AI)-assisted fundus images with other ophthalmic devices such as optical coherence tomography (OCT) and fundus fluorescence angiography (FFA) in the diagnosis of diabetic retinopathy and diabetic macular edema.

This study was conducted as a prospective study. Participants meeting eligibility criteria will be recruited from sites staffed by trained photographers. After assessing eligibility and obtaining informed consent, fundus photographs will be taken using a non-dilated fundus camera. And optical coherence tomography or fundus fluorescence angiography will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnostic for diabetes: Type 1 diabetes of a lest 5 years of evolution; or Type 2 diabetes;
2. Obtaining informed consent;
3. Patient age 18 or above.

Exclusion Criteria:

1. Patients under 18 years of age;
2. Failure to Obtain informed consent;
3. Presence of other retinal diseases;
4. A patient who has already undergone the treatment.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: It is planned to include 1,000 participants in the study, all of whom will undergo fundus photography, 500 additional patients will undergo fundus fluorescence angiography, and 500 additional patients will undergo optical coherence tomography.
  All participants met inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-07-10 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The accuracy | Baseline-Month 12
  Detection of DR accuracy using fundus photography, optical coherence tomography, and fundus fluorescence angiography

SECONDARY OUTCOMES:
The accuracy | Baseline-Month 12
  Detection of DME accuracy using fundus photography, optical coherence tomography, and fundus fluorescence angiography

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No